CLINICAL TRIAL: NCT05898399
Title: A Phase I/IIa, Open-label, Multi-center Study to Assess the Safety, Tolerability, Pharmacokinetics, and Preliminary Efficacy of the DNA Polymerase Theta Inhibitor ART6043 Administered Orally as Monotherapy and in Combination to Patients With Advanced or Metastatic Solid Tumors
Brief Title: Study of ART6043 in Advanced/Metastatic Solid Tumors Patients
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Artios Pharma Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ART6043C001
Record Dates: First submitted 2023-05-15; First posted 2023-06-12 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Advanced Solid Tumor; Metastatic Solid Tumor
Keywords: Metastatic Cancer; HER2-negative Breast Cancer; Poly (adenosine diphosphate ribose) polymerase (PARP) inhibitor (PARPi); Human epidermal growth factor receptor 2 negative (HER2-ve); Oral anticancer; Sensitivity to Polymerase Theta Inhibitor
MeSH Terms: conditions — Neoplasm Metastasis | interventions — olaparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Part A1 (ART6043 as monotherapy) (Experimental): Patients with advanced or metastatic cancer will receive ART6043 administered in 21-day cycles.
  Interventions: Drug: ART6043
- Part A2 (ART6043 in combination with olaparib) (Experimental): Patients with advanced or metastatic cancer and with PARPi as an appropriate treatment option will receive ART6043 in combination with olaparib twice daily (BID) in 21-day cycles.
  Interventions: Drug: ART6043; Drug: Olaparib
- Part B1 (ART6043 in combination with olaparib) (Experimental): Patients with g/sBRCA-m, HER2-ve locally advanced or metastatic breast cancer will be assigned to receive ART6043 in combination with olaparib.
  Interventions: Drug: ART6043; Drug: Olaparib
- Part B2 (ART6043 in combination with olaparib) (Experimental): Patients with g/sBRCA-m, HER2-ve locally advanced or metastatic breast cancer will be randomly assigned to receive ART6043 in combination with olaparib or olaparib alone.
  Interventions: Drug: ART6043; Drug: Olaparib

INTERVENTIONS:
Drug: ART6043 — ART6043 will be given orally.
Drug: Olaparib — Olaparib will be given orally.
  Arms: Part A2 (ART6043 in combination with olaparib); Part B1 (ART6043 in combination with olaparib); Part B2 (ART6043 in combination with olaparib)

SUMMARY:
This interventional study will evaluate the safety, tolerability, pharmacokinetics, and preliminary efficacy of ART6043 as monotherapy or in combination with olaparib.

DETAILED DESCRIPTION:
ART6043 is being developed as an oral anti-cancer agent in combination with a poly (adenosine diphosphate ribose) polymerase (PARP) inhibitor (PARPi) in patients with cancers that harbor defects in DNA repair.

The study will consist of two parts:

1. Part A (Dose-escalation phase): Part A will evaluate ART6043 as monotherapy (Part A1) in patients with advanced or metastatic cancer and in combination with olaparib (Part A2), in patients with advanced or metastatic cancer with genetic lesions that cause loss of function of known DNA Damage Response (DDR) genes. Olaparib is also referred as PARPi.
2. Part B (dose-expansion phase): To further confirm the safety of ART6043 in combination with olaparib (Part B1) and to assess initial effectiveness of ART6043 in combination compared to olaparib alone (Part B2) in patients with certain types of breast cancer.

Patients may continue to receive ART6043 and/or olaparib as long as they may be continuing to derive clinical benefit as assessed by the investigator and/or until disease progression, withdrawal of consent or until they experience unacceptable drug-related toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have discontinued all previous chemotherapeutic agents, non-hormonal targeted therapy, or investigational drugs for at least 21 days or 5 half-lives (not including palliative radiotherapy at focal sites), whichever is shorter. Endocrine and hormonal therapies for the treatment of cancer must have been discontinued (unless for the treatment of Prostate Cancer) at least 7 days before receiving study medication. Palliative radiotherapy must have completed prior to start of study treatment.
* Resolution of all toxicities of prior therapy or surgical procedures.
* Performance status of 0-2 on the Eastern Cooperative Oncology Group (ECOG) scale.
* Have adequate organ function.
* Patients of childbearing potential and patients with partners of childbearing potential are required to use highly effective contraception.
* Have an estimated life expectancy of ≥12 weeks, in the judgment of the investigator.

Inclusion Criteria specific to Part A1 (ART6043 as Monotherapy)

• Advanced or metastatic cancer. Tumors with genetic lesions known to cause loss of function of known DDR genes based on available pre-existing testing are encouraged.

Inclusion criteria specific to Part A2 (ART6043 in combination with olaparib)

* Advanced or metastatic cancer with genetic lesions known to cause loss of function of known DDR genes based on available, pre-existing testing.
* Patients for whom a PARPi is an appropriate treatment option. Patients may have received prior treatment with a PARPi.

Inclusion criteria specific to Part B (ART6043 in combination with olaparib or olaparib alone)

* Histologically or cytologically confirmed HER2-ve locally advanced or metastatic carcinoma of the breast.
* Documentation of a deleterious or suspected deleterious g/sBRCA mutation.
* No more than 3 prior chemotherapy-inclusive schedules (including antibody conjugates) for locally advanced and/or metastatic disease.
* Prior treatment with a taxane in the neoadjuvant, adjuvant, locally advanced, or metastatic setting unless medically contraindicated.
* Patients must have received no or ≤1 month of prior treatment with a PARPi.

Exclusion Criteria:

* Patients who are pregnant.
* Patients with Myelodysplastic syndrome (MDS)/Acute myeloid leukemia (AML) or with features suggestive of MDS/AML.
* Have ongoing interstitial lung disease or pneumonitis.
* Have any major gastrointestinal issues that could impact absorption of ART6043 or olaparib.
* Patients with brain metastases (patients with treated brain metastases could be eligible if follow-up brain imaging after central nervous system-directed therapy shows no evidence of progression).
* Have received a live vaccine within 30 days before the first dose of study treatment.
* Recent major surgery within 4 weeks prior to entry into the study.
* Have a significant bleeding disorder or vasculitis or had a Grade ≥3 bleeding episode within 12 weeks prior to enrollment.
* Have a history of allergy or hypersensitivity to study drug components.

Exclusion criteria specific to Part B

* First-line locally advanced and/or metastatic breast cancer with no prior adjuvant chemotherapy.
* Inflammatory breast cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2026-05-14 (Estimated); Study Completion 2026-12-14 (Estimated)

PRIMARY OUTCOMES:
Part A: Number of participants with Dose Limiting Toxicities (DLTs) | From first dose of study treatment until the end of Cycle 1 (each cycle is 21-days)
  Severity of adverse events as assessed by the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE) v5.0.
Part B1: Number of participants with adverse events | Screening (≤28 days) Until follow-up visit (90 days after discontinuation)] (up to 3.7 years)
  To assess the safety and tolerability of ART6043 given orally in combination with olaparib at the Recommended Phase II dose(s) [RP2D(s)].
Part B2: Progression free survival (PFS) | Until disease progression (Upto 3.7 years).
  PFS is defined as the time from randomization until objective disease progression as defined by Response evaluation criteria in solid tumors (RECIST) v1.1 or death by any cause in the absence of progression, regardless of whether the patient withdraws from study medication or receives another anti-cancer therapy prior to progression.

SECONDARY OUTCOMES:
Part B2: Number of participants with Adverse events | Screening (≤28 days) Until follow-up visit (90 days after discontinuation)] (up to 3.7 years)
  To assess the safety and tolerability of ART6043 given orally in combination with olaparib at the Recommended Phase II dose(s) [RP2D(s)].
Best overall response (BOR) | Screening (≤28 days) Until disease progression/recurrence (Upto 3.7 years)
  The best overall response is the best response (complete response [CR] or partial response [PR]) recorded from the date of randomization for each patient until the progression or censoring date in the absence of progression.
Objective Response Rate (ORR) | Screening (≤28 days) Until disease progression/recurrence (Upto 3.7 years)
  Objective Response Rate (ORR) is defined as the proportion of patients with a CR or PR to treatment according to RECIST v1.1.
Disease control rate (DCR) | Screening (≤28 days) Until disease progression (Upto 3.7 years)
  To assess preliminary signs of efficacy for ART6043 as monotherapy and in combination with olaparib.
Duration of response (DOR) | Screening (≤28 days) Until disease progression (Upto 3.7 years)
  The DOR will be defined for patients with a BOR of CR/PR (with a Prostate Cancer Working Group [3PCWG-3] response of non-PD/NE for patients with prostate cancer), as the time from the date of first documented response until date of documented progression (by RECIST v1.1 or PCWG-3) or death in the absence of disease progression.
Change in tumor size | Screening (≤28 days) Until disease progression (Upto 3.7 years)
  The best percentage change in tumor size from baseline will be determined for each patient, ie, the maximum reduction from baseline or the minimum increase from baseline in the absence of a reduction.
Change in level of cancer antigen 125 (CA-125) | Screening (≤28 days) Until follow-up visit (Upto 3.7 years)
  To assess preliminary signs of efficacy for ART6043 as monotherapy and in combination with olaparib.
Part A and B1: Progression free survival (PFS) | Screening (≤28 days) Until disease progression (Upto 3.7 years)
  The PFS is defined as the time from randomization until the earliest objective disease progression defined by RECIST v1.1 or PCWG-3 (for patients with prostate cancer in Arm 2) or death by any cause in the absence of progression, regardless of whether the patient withdraws from study medication or receives another anti-cancer therapy prior to progression.
Overall survival (OS) | Screening (≤28 days) Until overall survival follow-up (Upto 3.7 years)
  OS is defined as the time from the start of study treatment (Part A) or randomization (Part B) until death due to any cause.
Plasma concentration | Pre-dose Cycle 0 Days -2, -1 , Cycle 1 Days 1, 8, 15, 16, Cycle 2 Days 1, 8, 15, Cycle 3 Day 1 Upto 3.7 Years (Each Cycle is 21-Days)
  To determine the plasma concentration of ART6043 and its potential active metabolite ART7276 following both single and multiple oral dosing of ART6043 monotherapy and following multiple oral dosing of ART6043 in combination with olaparib. Also, to explore the effect of ART6043 on the Cmax of olaparib.
Half life (t1/2) | Pre-dose Cycle 0 Days -2, -1 , Cycle 1 Days 1, 8, 15, 16, Cycle 2 Days 1, 8, 15, Cycle 3 Day 1 Upto 3.7 Years (Each Cycle is 21-Days)
  To determine the t1/2 of ART6043 and its potential active metabolite ART7276 following both single and multiple oral dosing of ART6043 monotherapy and following multiple oral dosing of ART6043 in combination with olaparib. Also, to explore the effect of ART6043 on the t1/2 of olaparib.
Area under the plasma concentration-time curve from zero to infinity (AUC0-inf) | Pre-dose Cycle 0 Days -2, -1 , Cycle 1 Days 1, 8, 15, 16, Cycle 2 Days 1, 8, 15, Cycle 3 Day 1 Upto 3.7 Years (Each Cycle is 21-Days)
  To determine the AUC0-inf of ART6043 and its potential active metabolite ART7276 following both single and multiple oral dosing of ART6043 monotherapy and following multiple oral dosing of ART6043 in combination with olaparib. Also, to explore the effect of ART6043 on the AUC0-inf of olaparib.
Renal clearance | Cycle 0 Days -2, -1 (Each Cycle is 21-Days)
  To determine renal clearance of ART6043 and its potential active metabolite ART7276 following both single and multiple oral dosing of ART6043 monotherapy and following multiple oral dosing of ART6043 in combination with olaparib.
Percent of ART6043 excreted in urine | Cycle 0 Day -2 ((Each Cycle is 21-Days)
  To determine percent of ART6043 excreted in urine following single oral dosing of ART6043.
Cancer antigen 125 levels in pre-dose tumor samples | At Screening (≤28 days)
  To assess CA-125 levels in pre-dose tumor samples that may be predictive of the activity of ART6043.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - South Texas Accelerated Research Therapeutics (START) - Midwest, Grand Rapids, Michigan
  - Memorial Sloan-Kettering Cancer Center (MSKCC), New York, New York
  - Stephenson Cancer Center - Oncology, Oklahoma City, Oklahoma
  - Jefferson University Hospitals - Kimmel Cancer Center, Philadelphia, Pennsylvania
  - SCRI oncology partners, Nashville, Tennessee
  - Mary Crowley Cancer Center - Clinic, Dallas, Texas
  - The University of Texas - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No